CLINICAL TRIAL: NCT05239897
Title: Treatment of Postoperative Delirium With Continuous Theta Burst Stimulation: an Exploratory Study
Brief Title: Treatment of Postoperative Delirium With Continuous Theta Burst Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cTBStPOD
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- postoperative delirium (Experimental): We will use Confusion Assessment Method (CAM) to determine the incidence of postoperative delirium in participants twice per day. We will use the Memorial Delirium Assessment Scale(MDAS)and Mini-mental state examination(MMSE) to examine postoperative delirium severity.
  Interventions: Device: Continuous theta burst stimulation (cTBS)

INTERVENTIONS:
Device: Continuous theta burst stimulation (cTBS) — Patients assessed for postoperative delirium will be treated by consist of 600 pulses per session, delivered over the right dorsolateral prefrontal cortex at 80% of resting motor threshold (RMT). Every session cTBS consists of 50 Hz triplets of pulses delivered at 5 Hz for 40 seconds for a total of 600 pulses. Every set simulation includes 3 sessions.

SUMMARY:
To determine whether continuous theta burst stimulation can cure postoperative delirium in senior patients.

DETAILED DESCRIPTION:
Postoperative delirium(POD), a syndrome characterized by an acute change in attention, awareness and cognition, is one of the most common postoperative complications among elderly patients. Impaired neuronal network connectivity is likely one of the several neurobiological processes that contribute to POD pathogenesis. Recently, continuous theta burst stimulation (cTBS) was demonstrated to improve cognitive function in patients with mild cognitive impairment.Recent research suggests that cTBS has positive effect on improving the connectivity and reorganization of the brain network. Therefore, we plan to conduct an exploratory study in participants undergoing elective surgeries to determine whether cTBS can cure POD in this senior patient population.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60 to 80 years;
* Having delirium after elective surgery;
* Being able to complete cognitive assessment and confusion assessment methods (CAM);
* Willing to participate before surgery and being competent to provide informed consent.

Exclusion Criteria:

* Having brain tumor, stroke, or mental disorders (e.g., depression or dementia);
* Having contraindications of cTBS (e.g., head trauma, history of epilepsy or metal implants in the head or heart);
* Participating in other clinical studies.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Cure rate of POD after a single cTBS treatment | 7 days after surgery
  No POD was evaluated by CAM at 1 hour after a single cTBS treatment on the day of the first occurrence of POD and at any time point thereafter.

SECONDARY OUTCOMES:
Cure rate of POD after multiple cTBS treatments | 7 days after surgery
  No POD was evaluated by CAM at 1 hour after two or three cTBS treatments and at any time point thereafter.
Severity of postoperative delirium changed after each cTBS treatment | 7 days after surgery
  Severity of postoperative delirium on postoperative day 1 to 7 will be defined according to MDAS.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji hospital, School of medicine, Shanghai Jiaotong University, Pudong, Shanghai Municipality, China